CLINICAL TRIAL: NCT03061058
Title: An Open-label, Randomized, Phase III, Multicenter Clinical Trial Comparing the Efficacy and Safety of Individualized Intraperitoneal and System Chemotherapy Versus System Chemotherapy as First-line Chemotherapy for Advanced Gastric Cancer
Brief Title: Individualized Intraperitoneal and System Chemotherapy Versus System Chemotherapy as First-line Chemotherapy for AGC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yang Yang, Principal investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGC-PC
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Stomach Neoplasms; Chemotherapy Effect; Chemotherapeutic Toxicity
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Cisplatin; Irinotecan; Pemetrexed; S 1 (combination)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized Group (Experimental): mRNA levels of BRCA1, topoisomerase I (TOPO1), and thymidylate synthase (TS) were assessed in tumor tissue. Chemotherapeutic agents were selected based on the mRNA levels.
  Patients with high level BRCA1 will receive intraperitoneal docetaxel (15mg/m^2, d1, d15, q4w), intravenous docetaxel (30mg/m^2, d1, d15, q4w), and oral S-1 (40mg/m^2, d1-14, q4w).
  Patients with low level BRCA1 will receive intraperitoneal cisplatin (25mg/m^2, d1, d15, q4w), intravenous oxaliplatin (75mg/m^2, d1, d15, q4w), and oral S-1 (40mg/m^2, d1-14, q4w).
  Patients with middle level BRCA1 and high level TOPO1 will receive intraperitoneal irinotecan (45mg/m^2, d1, d15, q4w), intravenous docetaxel (90mg/m^2, d1, d15, q4w), and oral S-1 (40mg/m^2, d1-14, q4w).
  Patients with middle level BRCA1, low or middle level TOPO1, and low level TS will receive intraperitoneal pemetrexed (150mg/m^2, d1, q3w), and intravenous pemetrexed (350mg/m^2, d1, q3w).
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Cisplatin; Drug: Irinotecan; Drug: Pemetrexed; Drug: S1
- Control Group (Active Comparator): mRNA levels of BRCA1, TOPO1, and TS were assessed in tumor tissue for every enrolled patients.
  Patients in control group will receive intravenous docetaxel (45mg/m^2, d1, d15, q4w), and oral S-1 (40mg/m^2, d1-14, q4w).
  Interventions: Drug: Docetaxel; Drug: S1

INTERVENTIONS:
Drug: Docetaxel — intraperitoneal and/or intravenous
Drug: Oxaliplatin — intravenous
  Arms: Individualized Group
Drug: Cisplatin — intraperitoneal
  Arms: Individualized Group
Drug: Irinotecan — intraperitoneal and/or intravenous
  Arms: Individualized Group
Drug: Pemetrexed — intraperitoneal and/or intravenous
  Arms: Individualized Group
Drug: S1 — oral

SUMMARY:
Tumor messenger ribonucleic acid (mRNA) expression levels may have a promising role as potential predictive biomarkers for chemotherapy.

Peritoneal carcinomatosis appears to be the most common pattern of metastasis or recurrence and is associated with poor prognosis in gastric cancer patients. Intraperitoneal chemotherapy is widely accepted strategy in the treatment of peritoneal dissemination.

In this study, our aim is to evaluate the impact of individualized selection of chemotherapeutics and intraperitoneal combined with system chemotherapy on overall survival, disease free survival, response rate, and safety of advanced gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or metastatic disease, not amenable to curative therapy.
* Patients must have measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST, v1.1), assessed using imaging techniques (CT or MRI).
* Patients must have enough tumor tissue for mRNA expression test.
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to chemotherapy, postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential) and nonlactating, and men and women must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 6 months after therapy completed
* Eastern Cooperative Oncology Group (ECOG) Performance status 0, 1 or 2.
* Absolute neutrophil count (ANC) >=1,500/ul
* Platelets (PLT) >=75,000/ul
* Serum bilirubin <= 1.5 × upper limit of normal (ULN)
* Aspartate transaminase (AST) or alanine aminotransferase (ALT) <= 2.5 × ULN (or <= 5 × ULN in patients with liver metastases)
* Alkaline phosphatase <= 2.5 × ULN (or <= 5 × ULN in patients with liver metastases, or <= 10 × ULN in patients with bone but no liver metastases)
* Albumin >= 25 g/L.
* Creatinine clearance >= 60 mL/min.
* Life expectancy of at least 3 months.
* Signed informed consent.

Exclusion Criteria:

* Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study; the total dose of cisplatin should be less than 300mg/m^2).
* Patients with active (significant or uncontrolled) gastrointestinal bleeding.
* Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurological toxicity ≥ grade 2 NCI-CTCAE 4.0.
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
* History of documented congestive heart failure; angina pectoris requiring medication;evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
* Baseline left ventricular ejection fraction (LVEF) < 50% (measured by echocardiography or MUGA).
* Patients with dyspnoea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
* Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
* Clinically significant hearing abnormality.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* History or clinical evidence of brain metastases.
* Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
* Positive serum pregnancy test in women of childbearing potential.
* Received any investigational drug treatment within 4 weeks of start of study treatment.
* Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastatic site peripherally and patient recovered from any acute toxicity;prior adjuvant radiotherapy is allowed if complete at least 6 months ).
* Major surgery within 4 weeks of start of study treatment, without complete recovery.
* Patients with known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Known hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 1 year
  the follow-up visit of PFS will be performed every 6 weeks

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
Objective Response Rate | up to 24 weeks
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation
Adverse Events | up to 1 months
  participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Ma'anshan People's Hospital, Ma’anshan, Anhui
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Nanjing Gaochun People's Hospital, Nanjing, Jiangsu
  - Nanjing Lishui People's Hospital, Nanjing, Jiangsu
  - The Comprehensive Cancer Center of Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Suqian People's Hospital, Suqian, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: No